CLINICAL TRIAL: NCT00003156
Title: Evaluation of Topotecan in the Treatment of Persistent or Recurrent Carcinosarcoma (Mixed Mesodermal Tumors) of the Uterus
Brief Title: Topotecan in Treating Patients With Recurrent or Refractory Cancer of the Uterus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000065948; GOG-130D
Record Dates: First submitted 2000-11-06; First posted 2004-04-07 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2006-01

CONDITIONS: Sarcoma
Keywords: recurrent uterine sarcoma; uterine carcinosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Topotecan

INTERVENTIONS:
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of topotecan in treating patients with recurrent or refractory cancer of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the antitumor activity of topotecan in patients with recurrent or refractory carcinosarcoma of the uterus who have failed standard therapy. II. Determine the nature and degree of toxic effects of topotecan in these patients.

OUTLINE: Patients receive topotecan IV over 30 minutes daily for 5 days. Treatment repeats every 3 weeks for a minimum of 1 course in the absence of disease progression or unacceptable toxicity. Patients with complete response, partial response, or stable disease continue treatment for at least three courses. Patients are followed every 4 months for 2 years, every 6 months for 3 years, and then periodically thereafter until death.

PROJECTED ACCRUAL: Approximately 25-40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or refractory carcinosarcoma (mixed mesodermal tumors) of the uterus Measurable disease

PATIENT CHARACTERISTICS: Age: Not specified Performance Status: GOG 0-2 Life Expectancy: Not specified Hematopoietic: Platelet count at least 100,000/mm3 Absolute granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 3 times ULN Alkaline phosphatase no greater than 3 times ULN Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance greater than 20 mL/min Other: No invasive malignancies within the past 5 years except nonmelanomatous skin cancer No significant infection

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior biologic therapy Chemotherapy: At least 3 weeks since prior chemotherapy and recovered No prior topotecan or camptothecin therapy No more than 1 prior chemotherapy regimen (either single or combination chemotherapy) Endocrine therapy: At least 3 weeks since prior endocrine therapy Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: Prior surgery allowed and recovered

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-06; Primary Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Study Chair — Simmons Cancer Center
Locations (46):
- United States (45):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Sooner State, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Miller DS, Blessing JA, Schilder J, Munkarah A, Lee YC. Phase II evaluation of topotecan in carcinosarcoma of the uterus: a Gynecologic Oncology Group study. Gynecol Oncol. 2005 Aug;98(2):217-21. doi: 10.1016/j.ygyno.2005.05.015. PMID 15975641